CLINICAL TRIAL: NCT06511063
Title: Investigating the Feasibility of Repurposing HIV Antivirals in Adults With Long Covid
Brief Title: Antiviral Clinical Trial for Long Covid-19
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Yale University (Other); PolyBio Research Foundation (Other)
Responsible Party: Principal Investigator, David Putrino, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: STUDY-24-00088
Record Dates: First submitted 2024-07-16; First posted 2024-07-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Long Covid
Keywords: Long Covid; Antiviral; Truvada; Selzentry
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Maraviroc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Truvada (Tenofovir Disoproxil Fumarate, TDF/FTC, tenofovir disoproxil/emtricitabine) (Experimental): Participants will take 300mg tenofovir disoproxil fumarate/200 mg emtricitabine, once per day, and one placebo capsule per day, oral capsule for 90 days.
  Interventions: Drug: tenofovir disoproxil/emtricitabine; Drug: Placebo
- Selzentry (Experimental): Participants will take 300 mg of Selzentry, twice a day, oral capsule for 90 days.
  Interventions: Drug: Selzentry
- Placebo (Placebo Comparator): Participants will take a placebo, twice per day, oral capsule for 90 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tenofovir disoproxil/emtricitabine — Participants will take Truvada (TDF/FTC, tenofovir disoproxil/emtricitabine) for 90 days.
  Other Names: TDF/FTC; Truvada
  Arms: Truvada (Tenofovir Disoproxil Fumarate, TDF/FTC, tenofovir disoproxil/emtricitabine)
Drug: Selzentry — Participants will take Selzentry for 90 days.
  Arms: Selzentry
Drug: Placebo — Matching placebo.
  Arms: Placebo; Truvada (Tenofovir Disoproxil Fumarate, TDF/FTC, tenofovir disoproxil/emtricitabine)

SUMMARY:
The trial will test if two repurposed HIV antivirals can reduce symptom burden in adult participants with Long Covid compared to placebo. Viral infection and viral reactivation have been documented in Long Covid.

Participants will be randomly allocated to receive antivirals, Truvada (tenofovir disoproxil/emtricitabine, TDF/FTC, Group 1) or Selzentry (Group 2), or a placebo (pill) (Group 3), taken daily for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Any gender, aged 18+
* Diagnosed with:

  * Long Covid
  * Documented clinical history of confirmed or suspected acute SARS-CoV-2 infection a minimum of 6 months prior to contact with the study team
  * Formal diagnosis of Long Covid from a physician and a history of 6 months of Long COVID symptoms
* At least a six-month history of one of the following symptoms following SARS-CoV-2 infection:

  * headache, memory loss, insomnia, mood disturbance, chest pain, palpitations, shortness of breath, cough, muscle pains, joint pains, or GI upset] AND at least moderate fatigue (measured by Fatigue Severity Score) AND at least moderate post-exertional malaise (PEM) (measured by DePaul PEM screener)
* Participants who are willing and able to comply with all data collection, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Baseline EQ-VAS ≤70; EQ-VAS before the index infection ≥80 (this information is collected before randomization as part of the baseline survey).

Exclusion Criteria:

* Pre-existing conditions including, but not limited to:

  * Autoimmune conditions such as Chronic EBV, Multiple Sclerosis, Hashimoto's Disease, etc. which would impact the immunological profiling analysis.
  * A pre-2020 diagnosis of another Post-Acute Infectious Syndrome such as Chronic Lyme disease, Myalgic Encephalomyelitis/Chronic Fatigue Syndrome, etc.
  * Documented history of vaccine injury
  * Or any other chronic condition that has the potential to impact on immunological profiling, at the discretion of the research physician
* HIV+ status
* Current use of either Truvada or Selzentry
* Taking a medication, within 6 weeks, with known interactions with Truvada or Selzentry including but not limited to: Acyclovir, valacyclovir, adefovir, cabozantinib, carbamazepine, cidofovir, cladribine, cobicistat, diclofenac, multiple NSAIDs or chronic high dose NSAIDs, fosphenytoin or phenytoin, ganciclovir, valganciclovir, oxcarbazepine, phenobarbital, primidone, rifabutin, rifampin, rifapentine, sofosbuvir, tipranavir, or other drugs that significantly affect renal function
* Current treatment with drugs known to affect EBV replication, including but not limited to: Acyclovir, valacyclovir, ganciclovir, valganciclovir, famciclovir, teriflunomide, interferon
* Known allergic reactions to components of Truvada or Selzentry
* Febrile illness within the last 3 months of planned baseline evaluation
* Treatment with another investigational drug or other investigational intervention within 6 months of planned baseline evaluation
* Immunosuppressed individuals (transplant on antiviral prophylaxis and/or patients taking immunosuppressive medications such as steroids, etc.)
* Known medical history of active liver disease (other than nonalcoholic hepatic steatosis), including chronic or active hepatitis B or C infection, primary biliary cirrhosis, Child-Pugh Class B or C, or acute liver failure
* Receiving dialysis or have known renal impairment
* Any comorbidity requiring hospitalization and/or surgery within 7 days prior to study entry, or that is considered life threatening within days prior to study entry, as determined by the study team
* Other medical or psychiatric conditions, in the treating investigator's judgment, that makes the participant inappropriate for the study
* Unknown HIV status (subjects must have completed HIV antigen/antibody and viral load testing completed at the screening visit)
* Active or latent hepatitis B (subjects must have completed HBV serologies - HbsAg, anti-HBs, and anti-HBc - testing completed at the screening visit)
* Current symptoms of severe, progressive, or uncontrolled renal, hematologic, gastrointestinal, pulmonary, cardiac, or neurologic disease, or other medical conditions that, in the opinion of the investigator, might place the subject at unacceptable risk for participation in this study
* Creatinine clearance (CrCl) <75mL/min, as calculated by the Cockcroft-Gault equation
* Any history of bone fractures not explained by trauma
* Confirmed Grade 2 or greater hypophosphatemia
* Any Grade 2 or greater toxicity on screening tests and assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
EuroQol 5-Dimension 5-Level (EQ-5D-5L) Visual Analogue Scale | at Screening, Day 60, Day 90, and Day 180
  The EQ-5D-5L is a standardized measure of health status that consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each with 5 levels of severity, and a visual analogue scale (VAS) where individuals rate their overall health from 0 (worst imaginable health) to 100 (best imaginable health).

SECONDARY OUTCOMES:
The EuroQol Five-Dimensional Health Questionnaire (EQ-5D-5L) | at Screening, Day 60, Day 90, and Day 180
  The EQ-5D-5L is a validated, standardized, generic instrument that is a preference-based health- related quality of life questionnaire. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate their health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. Full scale from 5 to 25, with higher score indicating poorer health outcomes.
Patient-Reported Outcomes Measurement Information System 29 (PROMIS-29) | at Screening, Day 60, Day 90, and Day 180
  The PROMIS-29 v2.0 profile assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain. The values of all item responses are averaged to generate subscores for each dimension. From these subscores, a global physical health score and a global mental health score are generated. The scores are translated into T-scores according to a reference population with a mean of 50 and a standard deviation of 10.
General Symptom Questionnaire (GSQ-30) | at Screening, Day 60, Day 90, and Day 180
  The General Symptom Questionnaire-30 (GSQ-30) is a valid and reliable instrument to assess symptom burden among patients with acute and post-treatment. The GSQ-30 total score ranges from 0 to 120, with higher scores indicating a greater symptom burden.
Patient Health Questionnaire (PHQ-9) | at Screening, Day 60, Day 90, and Day 180
  The PHQ-9 is a series of questions assessing presence and severity of depression symptoms. It evaluates each of the DSM-IV depression criteria and scores the responses from 0 ("Not at all") to 3 ("Nearly every day"). PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively. Full scale from 0-27, with higher score indicating more severe symptoms.
Generalized Anxiety Disorder (GAD-7) | at Screening, Day 60, Day 90, and Day 180
  The GAD-7 is a 7-item scale developed and validated to identify generalized anxiety disorder and its severity. It assesses the frequency of 7 anxiety symptoms and scores the responses from 0 ("Not at all") to 3 ("Nearly every day"). Total scores of 5, 10, and 15 correspond to mild, moderate, and severe generalized anxiety disorder, respectively. Full scale from 0-21, with higher score indicating more symptoms.
Neuro-QoL™ v2.0 Cognitive Function-Short Form | at Screening, Day 60, Day 90, and Day 180
  The Neuro-QoL Cognitive Function v2.0 short form assesses perceived difficulties in cognitive abilities, including memory, attention, decision making, planning, organizing, calculating, remembering, and learning. The short form consists of 8 questions assessed on a 5-point Likert scale, resulting in a raw score range of 8 to 40. A raw score is then converted to a T-score using conversion tables. Scores 0.5 - 1.0 SD worse than the mean (T-score 40-45) = mild symptoms/impairment. Scores 1.0 - 2.0 SD worse than the mean (T-score 30-40) = moderate symptoms/impairment. Scores 2.0 SD or more worse than the mean (T-score below 30) = severe symptoms/impairment.
Single-item Sleep Quality Scale (SQS) | at Screening, Day 60, Day 90, and Day 180
  The SQS is a visual analog scale that instructs respondents to rate their overall quality of sleep over a 7-day recall period from 0 to 10. Scores of 0, 1, 4, 7, and 10 correspond to terrible, poor, fair, good, and excellent, respectively. Higher scores indicate better sleep quality.
Fatigue Severity Scale (FSS) | at Screening, Day 60, Day 90, and Day 180
  The Fatigue Severity Scale (FSS) uses a 7-point scale (1-7) to assess fatigue, with higher scores indicating greater severity, and a total score ranging from 9 to 63. Higher scores indicate more severe fatigue.
Fatigue Visual Analogue Scale (F-VAS) | at Screening, Day 60, Day 90, and Day 180
  The F-VAS consists of 18 items related to fatigue and energy in a visual analogue scale from 0 to 100. A higher score indicates more fatigue.
DePaul Post-Exertional Malaise Questionnaire (DSQ) | at Screening, Day 60, Day 90, and Day 180
  The DSQ is designed to evaluate 54 classic ME/CFS symptoms, including fatigue, post-exertional malaise, sleep, pain, neurological/cognitive impairments, and autonomic, neuroendocrine, and immune symptoms. Each symptom's frequency and intensity are rated on a 5-point scale (0-4). Frequency and severity scores are multiplied by 25, added together, and then divided by 2 to create a composite frequency/severity score for each symptom. These scores range from 0 to 100, with higher scores indicating a greater symptom burden.
Composite Autonomic Symptom Score 31(COMPASS-31) | at Screening, Day 60, Day 90, and Day 180
  The COMPASS-31 is a 31-question self-assessment instrument of autonomic symptoms and function that is up-to-date, broadly applicable, easy to administer in a short amount of time, and based on a scientific approach. The total score ranges from 0 to 100, with higher scores indicating greater autonomic dysfunction.
Pain Visual Analogue Scale (P-VAS) | at Screening, Day 60, Day 90, and Day 180
  Using a visual analogue scale, patients mark a point on a line representing a continuum from "no pain" to "worst pain," with scores ranging from 0 to 100, where higher scores indicate greater pain.

CONTACTS AND LOCATIONS:
Overall Officials: David Putrino, PhD, PT, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- The Cohen Center for Recovery from Complex Chronic Illnesses (CoRE), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No